CLINICAL TRIAL: NCT04439799
Title: A Comparison of Side Effects in Hypogonadal Men Treated With Natesto Versus Testosterone Injections: A Phase IV, Prospective, Randomized, Non-Blinded, Multi-Institutional Study
Brief Title: A Comparison of Side Effects in Hypogonadal Men Treated With Natesto Versus Testosterone Injections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Acerus Pharmaceuticals Corporation (Industry)
Responsible Party: Principal Investigator, Ranjith Ramasamy, MD, Director of Male Fertility and Andrology, University of Miami, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200201
Record Dates: First submitted 2020-05-25; First posted 2020-06-19 (Actual); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: Hypogonadism, Male
Keywords: Low T
MeSH Terms: conditions — Eunuchism | interventions — testosterone 17 beta-cypionate; Natesto

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testosterone Cypionate Group (Active Comparator): Participants in this group will receive the intramuscular Testosterone Cypionate intervention for four months
  Interventions: Drug: Testosterone Cypionate 200 Mg/ML
- Natesto Group (Active Comparator): Participants in this group will receive the intranasal testosterone (Natesto) intervention for four months.
  Interventions: Drug: Intranasal Testosterone

INTERVENTIONS:
Drug: Testosterone Cypionate 200 Mg/ML — Participants in this group will receive intramuscular testosterone cypionate injections of 1 cc (200mg) once every 14 days for four months.
  Arms: Testosterone Cypionate Group
Drug: Intranasal Testosterone — Participant in this group will receive Intranasal testosterone administered using a multi-dose dispenser, as two or three daily doses (5.5 mg per nostril, 11.0 mg single dose) for 4 consecutive months,
  Other Names: Natesto
  Arms: Natesto Group

SUMMARY:
The purpose of this study is to evaluate changes in vascular parameters and the prevalence of side effects in subjects receiving 1 cc (200mg) every 2 weeks intramuscular (IM) of Testosterone Cypionate versus subjects receiving 11mg three times daily (TID) Natesto to participant with clinical hypogonadism.

DETAILED DESCRIPTION:
Administration of exogenous testosterone as efficacious treatment for male hypogonadism has been part of medical practice for more than 50 years. Testosterone replacement therapy (TRT) is becoming more widely available and has seen a greater than three-fold increase in use in men 40 years and older. Current delivery systems of TRT include transdermal gels and patches, intranasal gels (currently marketed as Natesto), injection therapy, and long acting subcutaneous pellets.

Natesto is a short-acting formulation of testosterone delivered intranasally to men diagnosed with low T. This has the potential to avoid side effects related to TRT that are commonly seen with other delivery methods, namely polycythemia, acne, male-pattern hair loss, azoospermia and hyperestrogenemia.

Testosterone Cypionate injections are the most common form of TRT in the USA. Testosterone Cypionate has many reported side effects, the most common being polycythemia, gynecomastia, hair loss, acne, decreased spermatogenesis, and testicular atrophy. In a multicenter retrospective study, it has been shown that the prevalence of polycythemia in men on testosterone replacement (injections) was 11.2%. In this study, we will compare hematocrit changes caused by treatment with Testosterone Cypionate and Natesto in a parallel arm, randomized study. To date, there have been no direct head-to-haed comparisons of these formulations.

We hypothesize that the short-acting pharmacokinetics of Natesto more closely resembles the natural pulsatility of testosterone and therefore can avoid side effects traditionally seen in long-acting, exogenous testosterone formulations

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign and date the study consent form(s), which have been approved by an Institutional Review Board (IRB). Written consent must be obtained prior to the initiation of any study procedures.
2. Documented diagnosis of primary hypogonadism (congenital or acquired) or hypogonadotropic hypogonadism (congenital or acquired).
3. Serum total testosterone < 300 ng/dL on 2 measurements
4. Naïve to androgen replacement or has discontinued current treatment and completed a washout of 4 months following androgen treatment.
5. Men deemed to be candidates for TRT based on the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG).

Exclusion Criteria:

1. History of significant sensitivity or allergy to androgens, or product excipients.
2. Clinically significant findings in the pre-study examinations including abnormal breast examination requiring follow-up, abnormal ECG.
3. Abnormal prostate digital rectal examination (DRE) with palpable nodule(s)
4. Body mass index (BMI) ≥ 40 kg/m2.
5. Clinically significant abnormal laboratory value, in the opinion of the investigator, in serum chemistry, hematology, or urinalysis including but not limited to:

   1. Baseline hemoglobin > 16 g/dL or Hematocrit (HCT) 48%
   2. Prostate Specific Antigen (PSA) > 4 ng/mL
6. History of seizures or convulsions, including febrile, alcohol or drug withdrawal seizures.
7. History of any clinically significant illness, infection, or surgical procedure within 4 weeks prior to study drug administration.
8. History of stroke or myocardial infarction within the past 5 years.
9. History of, or current or suspected, prostate or breast cancer.
10. History of diagnosed, severe, untreated, obstructive sleep apnea.
11. History of abuse of alcohol or any drug substance in the opinion of the investigator within the previous 2 years.
12. Donation or loss of 550 mL or more blood volume (including plasmapheresis) or receipt of a transfusion of any blood product within 12 weeks prior to the start of treatment.
13. Inadequate venous access for collection of serial blood samples required for pharmacokinetic profiles.
14. Receipt of any subcutaneous testosterone pellets within the last 6 months.
15. Inability to understand and provide written informed consent for the study.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranjith Ramasamy, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corona G, Rastrelli G, Maggi M. Diagnosis and treatment of late-onset hypogonadism: systematic review and meta-analysis of TRT outcomes. Best Pract Res Clin Endocrinol Metab. 2013 Aug;27(4):557-79. doi: 10.1016/j.beem.2013.05.002. Epub 2013 Jul 5. PMID 24054931
- [Background] Haring R, Volzke H, Steveling A, Krebs A, Felix SB, Schofl C, Dorr M, Nauck M, Wallaschofski H. Low serum testosterone levels are associated with increased risk of mortality in a population-based cohort of men aged 20-79. Eur Heart J. 2010 Jun;31(12):1494-501. doi: 10.1093/eurheartj/ehq009. Epub 2010 Feb 17. PMID 20164245
- [Background] Walker WH. Testosterone signaling and the regulation of spermatogenesis. Spermatogenesis. 2011 Apr;1(2):116-120. doi: 10.4161/spmg.1.2.16956. PMID 22319659
- [Background] Katznelson L, Finkelstein JS, Schoenfeld DA, Rosenthal DI, Anderson EJ, Klibanski A. Increase in bone density and lean body mass during testosterone administration in men with acquired hypogonadism. J Clin Endocrinol Metab. 1996 Dec;81(12):4358-65. doi: 10.1210/jcem.81.12.8954042.
- [Background] Finkelstein JS, Klibanski A, Neer RM, Greenspan SL, Rosenthal DI, Crowley WF Jr. Osteoporosis in men with idiopathic hypogonadotropic hypogonadism. Ann Intern Med. 1987 Mar;106(3):354-61. doi: 10.7326/0003-4819-106-3-. PMID 3544993
- [Background] Jockenhovel F, Vogel E, Reinhardt W, Reinwein D. Effects of various modes of androgen substitution therapy on erythropoiesis. Eur J Med Res. 1997 Jul 28;2(7):293-8. PMID 9233903
- [Background] Behre HM, Bohmeyer J, Nieschlag E. Prostate volume in testosterone-treated and untreated hypogonadal men in comparison to age-matched normal controls. Clin Endocrinol (Oxf). 1994 Mar;40(3):341-9. doi: 10.1111/j.1365-2265.1994.tb03929.x. PMID 7514512
- [Background] Davidson JM, Camargo CA, Smith ER. Effects of androgen on sexual behavior in hypogonadal men. J Clin Endocrinol Metab. 1979 Jun;48(6):955-8. doi: 10.1210/jcem-48-6-955. PMID 447801
- [Background] Snyder PJ, Peachey H, Berlin JA, Hannoush P, Haddad G, Dlewati A, Santanna J, Loh L, Lenrow DA, Holmes JH, Kapoor SC, Atkinson LE, Strom BL. Effects of testosterone replacement in hypogonadal men. J Clin Endocrinol Metab. 2000 Aug;85(8):2670-7. doi: 10.1210/jcem.85.8.6731. PMID 10946864
- [Background] Baillargeon J, Urban RJ, Ottenbacher KJ, Pierson KS, Goodwin JS. Trends in androgen prescribing in the United States, 2001 to 2011. JAMA Intern Med. 2013 Aug 12;173(15):1465-6. doi: 10.1001/jamainternmed.2013.6895. No abstract available. PMID 23939517
- [Background] Ullah MI, Riche DM, Koch CA. Transdermal testosterone replacement therapy in men. Drug Des Devel Ther. 2014 Jan 9;8:101-12. doi: 10.2147/DDDT.S43475. eCollection 2014. PMID 24470750
- [Derived] Rivero MJ, Ory J, Diaz P, Thirumavalavan N, Han S, Reis IM, Ramasamy R. Comparison of Hematocrit Change in Testosterone-deficient Men Treated With Intranasal Testosterone Gel vs Intramuscular Testosterone Cypionate: A Randomized Clinical Trial. J Urol. 2023 Jul;210(1):162-170. doi: 10.1097/JU.0000000000003487. Epub 2023 May 1. PMID 37126399

RESULTS

PARTICIPANT FLOW:
Groups:
- Natesto Group: Participants in this group will receive the intranasal testosterone (Natesto) intervention for four months.
  Intranasal Testosterone: Participant in this group will receive Intranasal testosterone administered using a multi-dose dispenser, as three daily doses (5.5 mg per nostril, 11.0 mg single dose) for four consecutive months,
Period: Overall Study
Arm/Group | Testosterone Cypionate Group | Natesto Group
Started | 41 | 40
Completed | 31 | 23
Not Completed | 10 | 17
Not completed — Lost to Follow-up | 6 | 6
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Adverse Event | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone Cypionate Group | Natesto Group | Total
Number analyzed (Participants) | 41 | 40 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.46 (11.86) | 48.2 (10.89) | 48.33 (11.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 41 | 40 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 22 | 51
  Not Hispanic or Latino | 12 | 18 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 9 | 9
  White | 40 | 29 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Hematocrit (Hct) Levels.
Description: Changes in serum Hematocrit levels will be assessed in percentage
Time Frame: Baseline to 4 months
Measure: Mean (95% Confidence Interval); unit: percentage of hematocrit
Arm/Group | Testosterone Cypionate Group | Natesto Group
Number analyzed (Participants) | 31 | 23
percentage of hematocrit | 3.0 [2.8 to 5] | -0.6 [-1.5 to 0.4]

2. Secondary Outcome: Change in Hormone Levels
Description: Change in serum hormone levels including Testosterone, 17-Hydroxyprogesterone (17-OHP) assessed in ng/dL.
Time Frame: Baseline to 4 months
Population: In the Natesto group, three participants group did not have Testosterone labs collected and four did not have 17-OHP laboratory tests collected due to protocol non-compliance. in the Testosterone Cypionate group, Nine group did not have 17-OHP labs collected due to protocol non-compliance.
Measure: Mean (95% Confidence Interval); unit: ng/dL
Arm/Group | Testosterone Cypionate Group | Natesto Group
Number analyzed (Participants) | 31 | 20
ng/dL
  Testosterone | 511 [373 to 650] | 283 [149 to 417]
  17-OHP: number analyzed (Participants) | 22 | 19
  17-OHP | -39.8 [-53.1 to -26.5] | -8.8 [-24.4 to 6.7]

3. Secondary Outcome: Change in PSA Levels
Description: Change in serum Prostate Specific Antigen (PSA) levels will be assessed in ng/mL.
Time Frame: Baseline to 4 months
Population: Six participants in the Testosterone Cypionate group did not have PSA laboratory tests performed due to protocol non-compliance. Six participants in the Natesto group did not have PSA laboratory tests performed due to protocol non-compliance.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Testosterone Cypionate Group | Natesto Group
Number analyzed (Participants) | 25 | 17
ng/mL | 0.6 [-0.02 to 1.23] | 0.05 [-0.22 to 0.32]

4. Secondary Outcome: Change in Estradiol Levels
Description: Change in serum estradiol levels will be assessed in pg/mL.
Time Frame: Baseline to 4 months
Population: In the Testosterone Cypionate group, seven participants did not have estradiol laboratory tests performed due to protocol non-compliance. in the Natesto group three participants did not have estradiol laboratory tests performed due to protocol non-compliance.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Testosterone Cypionate Group | Natesto Group
Number analyzed (Participants) | 24 | 20
pg/mL | 22.9 [11 to 34.8] | 1.1 [-5.7 to 7.8]

5. Secondary Outcome: Changes in IIEF-6 Score
Description: The International Index of Erectile Function (IIEF)-6 is a 6-item subdomain self-evaluation questionnaire of erectile function. Each item is scored from 0-5 with the total score ranging from 0-30 with the higher score indicating better erectile function.
Time Frame: Baseline to 4 months
Population: In the Testosterone Cypionate group, fourteen participants did not complete the IIEF-6 questionnaire due to protocol non-compliance. In the Natesto group thirteen participants did not complete the IIEF-6 questionnaire due to protocol non-compliance.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Testosterone Cypionate Group | Natesto Group
Number analyzed (Participants) | 17 | 10
score on a scale | 4.8 [1.1 to 8.5] | 0.2 [-3.6 to 4]

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Testosterone Cypionate Group | Natesto Group
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/40
Other Adverse Events (participants affected / at risk) | 2/41 | 5/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Cypionate Group (N=41) | Natesto Group (N=40)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Labyrithitis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Generalized Edema (General disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT04439799/Prot_SAP_000.pdf